CLINICAL TRIAL: NCT05228457
Title: Intensive TMS for Rapid Relief of Bipolar Depression Symptoms
Brief Title: Intensive TMS for Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Yvette Sheline, McLure Professor of Radiology, Neurology and Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 850359
Record Dates: First submitted 2022-01-13; First posted 2022-02-08 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Bipolar Depression; Treatment Resistant Depression
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active Transcranial Magnetic Stimulation (Active Comparator): Active Intensive iTBS involves intermittent theta-burst stimulation (iTBS), a patterned form of repetitive transcranial magnetic stimulation (rTMS) over the left dorsal lateral prefrontal cortex (L-DLPFC).
  Interventions: Device: Intensive intermittent theta-burst stimulation (iTBS)
- Sham Transcranial Magnetic Stimulation (Sham Comparator): Sham Intensive iTBS involves using the coil's electric stimulation functionality that allows for the delivery of a brief electric pulse to the scalp simultaneous to the TMS pulse, which mimics the scalp sensation from active stimulation.
  Interventions: Device: Intensive intermittent theta-burst stimulation (iTBS)

INTERVENTIONS:
Device: Intensive intermittent theta-burst stimulation (iTBS) — Intensive iTBS is intermittent theta-burst stimulation (iTBS), a patterned form of repetitive transcranial magnetic stimulation (rTMS) over a specific brain region.

SUMMARY:
The research study is being conducted to test whether using high dose spaced theta-burst rTMS (a form of transcranial magnetic stimulation) produces a significant reduction in depressive symptoms compared with sham. This project will recruit patients aged 18-70 with symptoms of bipolar depression who have failed (or not shown signs of improvement) after at least two prior treatments.

DETAILED DESCRIPTION:
The research study is being conducted to test whether using high dose spaced theta-burst rTMS (a form of transcranial magnetic stimulation) produces a significant reduction in depressive symptoms compared with sham. This project will recruit patients aged 18-70 with symptoms of bipolar depression who have failed (or not shown signs of improvement) after at least two prior treatments. The null hypothesis is that there will be no difference in reductions in depressive symptoms by the end of a five-day treatment period. The alternative hypothesis is that, compared with sham, active TMS will result in a greater reduction in depressive symptoms by the end of the treatment period. Participants will be randomly assigned to active or sham conditions: 50% to active and 50% to sham.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar depression (BP I and BP II) by Diagnostic and Statistical Manual 5 (DSM 5) criteria
* Age 18-70
* Right or left handed
* All genders
* Treatment resistant depression, as in they must have treatment resistant depression with 2 or more prior antidepressant trials that have failed to produce a response (> 50% reduction in symptoms) using ATHF criteria
* Able to provide informed consent to participate in the study
* Must be on a stable medication regimen, requiring at least one mood stabilizer
* Depression severity as represented by scoring at least 20 on Montgomery-Asberg Depression Rating Scale (MADRS)

Exclusion Criteria:

* No current substance abuse disorder for the past 6 months (previous substance abuse not exclusionary)
* Any psychotic disorder or current active psychotic symptoms (personality disorders not exclusionary unless in the opinion of the referring psychiatrist it would jeopardize participation)
* No dementia or other major neurological disorders
* Not having depression as primary disorder
* No major medical illness, for example metastatic cancer, end stage renal disease
* Not able to verify contact information. Participants must be able to follow through with the study & must have verified contact information and at least one verified contact
* Pregnancy. While there are no known risks to a fetus this is a new use of TMS, which has not been tested, thus pregnancy is exclusionary
* Score on Young Mania Rating Scale (YMRS) greater than 12 (patients with mixed features have been shown not to respond well to TMS treatment)
* Rapid cycling Bipolar illness (patients with > 4 mood episodes within the past year will be excluded, as they have a higher risk of switch to mania)
* Any implants, conditions, or contraindications that would be deemed unsafe for TMS or MRI
* Currently using benzodiazepines (such as lorazepam) with a dose >1 mg per day or equivalent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Sheline, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Neuromodulation in Depression and Stress, University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Sheline YI, Makhoul W, Batzdorf AS, Nitchie FJ, Lynch KG, Cash R, Balderston NL. Accelerated Intermittent Theta-Burst Stimulation and Treatment-Refractory Bipolar Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2024 Sep 1;81(9):936-941. doi: 10.1001/jamapsychiatry.2024.1787. PMID 38985492

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-four participants were assessed for eligibility. Of these, eight did not meet the inclusion criteria and were excluded: three participants displayed manic symptoms at screening, four did not meet the criteria for major depression, and one did not meet the criteria for bipolar disorder.
Groups:
- Active Transcranial Magnetic Stimulation: Active Intensive iTBS involves intermittent theta-burst stimulation (iTBS), a patterned form of repetitive transcranial magnetic stimulation (rTMS) over the left dorsal lateral prefrontal cortex (L-DLPFC).
  Intensive intermittent theta-burst stimulation (iTBS): Intensive iTBS is intermittent theta-burst stimulation (iTBS), a patterned form of repetitive transcranial magnetic stimulation (rTMS) over a specific brain region.
  Active TMS was administered every day for five days over the course of nine hours. Every hour, the participant received nine minutes of TMS treatment for a total of 10 sessions a day.
- Sham Transcranial Magnetic Stimulation: Sham Intensive iTBS involves using the coil's electric stimulation functionality that allows for the delivery of a brief electric pulse to the scalp simultaneous to the TMS pulse, which mimics the scalp sensation from active stimulation.
  Intensive intermittent theta-burst stimulation (iTBS): Intensive iTBS is intermittent theta-burst stimulation (iTBS), a patterned form of repetitive transcranial magnetic stimulation (rTMS) over a specific brain region.
  Sham TMS was administered every day for five days over the course of nine hours. Every hour, the participant received nine minutes of sham TMS treatment and total of 10 sessions a day.
Period: Overall Study
Arm/Group | Active Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Started | 13 | 13
Completed | 12 | 12
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Thirteen participants were randomized to receive active TMS, and thirteen were randomized to receive sham TMS. One participant from each group withdrew from the study due to time commitment constraints, resulting in their exclusion from the analysis. Therefore, twelve participants from each group completed the study and were included in the final analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Thirteen participants were randomized to receive active TMS, and thirteen were randomized to receive sham TMS. One participant from each group withdrew from the study due to time commitment constraints, resulting in their exclusion from the analysis. Therefore, twelve participants from each group completed the study and were included in the final analysis
  years
    number analyzed (Participants) | 12 | 12 | 24
    (all) | 45 (14.7) | 44 (19.2) | 44.5 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Thirteen participants were randomized to receive active TMS, and thirteen were randomized to receive sham TMS. One participant from each group withdrew from the study due to time commitment constraints, resulting in their exclusion from the analysis. Therefore, twelve participants from each group completed the study and were included in the final analysis.
  Participants
    number analyzed (Participants) | 12 | 12 | 24
    Female | 6 | 6 | 12
    Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Thirteen participants were randomized to receive active TMS, and thirteen were randomized to receive sham TMS. One participant from each group withdrew from the study due to time commitment constraints, resulting in their exclusion from the analysis. Therefore, twelve participants from each group completed the study and were included in the final analysis
  Participants
    number analyzed (Participants) | 12 | 12 | 24
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 2 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 1 | 3
    White | 9 | 9 | 18
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Efficacy of High Dose Spaced Theta Burst (HDS-TBS)
Description: The primary outcome will be based on the set of repeated Montgomery Asberg Depression scores (10 items rated on a 0-6 scale, 0-60 possible score range, with higher scores indicating greater depressive symptomology), obtained at baseline, on each of the five treatment days and post TMS.
Time Frame: Through study completion, approximately 1 week
Population: Thirteen participants (age between 18-70)were randomized to receive active TMS, and thirteen were randomized to receive sham TMS. One participant from each group withdrew from the study due to time commitment constraints, resulting in their exclusion from the analysis. Therefore, twelve participants from each group completed the study and were included in the final analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active Transcranial Magnetic Stimulation: Active Intensive iTBS involves intermittent theta-burst stimulation (iTBS), a patterned form of repetitive transcranial magnetic stimulation (rTMS) over the left dorsal lateral prefrontal cortex (L-DLPFC).
  Intensive intermittent theta-burst stimulation (iTBS): Intensive iTBS is intermittent theta-burst stimulation (iTBS), a patterned form of repetitive transcranial magnetic stimulation (rTMS) over a specific brain region.
  Active TMS was administered every day for five days over the course of nine hours. Every hour, the participant received nine minutes of sham TMS treatment and total of 10 sessions a day.
Arm/Group | Active Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 12 | 12
score on a scale
  baseline | 30.4 (4.81) | 28 (5.41)
  treatment end | 10.5 (6.76) | 25.3 (6.74)
  Day 1 | 26.7 (2.27) | 26.8 (6.19)
  Day 2 | 20.3 (6.27) | 25.7 (5.55)
  Day 3 | 16.3 (7.65) | 24.3 (5.94)
  Day 4 | 11.3 (7.23) | 24.8 (4.81)
  Day 5 | 10.2 (7.56) | 25.3 (6.74)
Statistical Analysis 1: Comparison: Active Transcranial Magnetic Stimulation vs Sham Transcranial Magnetic Stimulation; Test type: Superiority — 13 participants were randomized to receive active TMS, and 13 were randomized to receive sham TMS. 1 participant from each group withdrew, resulting in their exclusion from the analysis. Therefore, 24 participants were randomized to active (n = 12) or sham (n = 12) aiTBS groups. The analysis examined MADRS scores measured at baseline and post-treatment. A priori hypotheses were that active aiTBS would demonstrate measurable differences in MADRS scores compared to the sham group; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -14.8, 95% CI 2-sided [-19.94 to -9.56] — The primary outcome was the between-group (Active vs Sham) difference in MADRS scores at the end of the treatment period. Results, including mean scores, standard deviations, confidence intervals, and p-value for the between-group comparisons

2. Secondary Outcome: Relationship Between Change in Brain Resting State Functional Connectivity and Treatment Effects
Description: The secondary outcome will be the change in the correlation between the dorsolateral prefrontal cortex (DLPFC) and the subgenual anterior cingulate cortex (sgACC) with the Montgomery-Åsberg Depression Rating Scale (MADRS), as assessed through MRI scans conducted at baseline and post-stimulation. Additionally, the change in the correlation within the entire Default Mode Network (DMN) intraconnectivity and MADRS will be measured for both groups (Active vs. Sham). The correlation is measured on a scale from -1 to +1, where -1 indicates the highest negative anticorrelation, +1 represents the highest positive correlation, and 0 signifies no correlation. MADRS is used to assess the clinical effect.
Time Frame: Upon study completion, approximately 1 week
Population: Thirteen participants (age between 18-70) were randomized to receive active TMS, and thirteen were randomized to receive sham TMS. One participant from each group withdrew from the study due to time commitment constraints, resulting in their exclusion from the analysis. Therefore, twelve participants from each group completed the study and were included in the final analysis.
Measure: Mean (Full Range); unit: correlation coefficient
Arm/Group | Active Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
Number analyzed (Participants) | 12 | 12
correlation coefficient
  Correlation between connectivity between (DLPFC) vs (sgACC) and MADRS. | -0.63 [-1 to 1] | 0.33 [-1 to 1]
  Correlation between the whole Default Mode Network (DMN) intraconnectivity and MADRS | 0.15 [-1 to 1] | -0.43 [-1 to 1]
Statistical Analysis 1: Comparison: Active Transcranial Magnetic Stimulation; Z-transformed Pearson's r values of average voxel-wise connectivity within the DMN; Test type: Superiority; p = 0.04, t-test, 2 sided; Z-transformed Pearson's r values = -0.014

ADVERSE EVENTS:
Time Frame: For each participant, adverse events were recorded from baseline to the end of participation, typically about 6 weeks. This randomized clinical trial was conducted from March 2022 to February 2024, with all adverse event data collected throughout this period.
Arm/Group | Active Transcranial Magnetic Stimulation | Sham Transcranial Magnetic Stimulation
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 6/13 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Transcranial Magnetic Stimulation (N=13) | Sham Transcranial Magnetic Stimulation (N=13)
Headache (Nervous system disorders) | 5 (5) | 2 (2) — A mild headache occurred after the participant received TMS. It was of low intensity and resolved within a few hours without any intervention.
dizziness (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT05228457/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT05228457/ICF_002.pdf